CLINICAL TRIAL: NCT03789201
Title: Exploring the Relationship Between Brain Asymmetry and Attention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 190036; 19-N-0036
Record Dates: First submitted 2018-12-27; First posted 2018-12-28 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10-24

CONDITIONS: Normal Physiology
Keywords: TMS-Evoked Potential; TMS; fMRI; Behavior; Electroencephalogram (EEG)
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Volunteers (Experimental): thematic permission to use non-invasive techniques regarded as having minimal risk in healthy individuals, such as, MRI, EEG, EMG, low-frequency stimulation (= 1 Hz), electrical stimulation of the skin to mimic the somatosensory artifact of TMS, and behavioral tests
  Interventions: Device: TMS EEG; Device: TMS fMRI

INTERVENTIONS:
Device: TMS EEG — attempt to use TMS EEG to measure connectivity between cortical areas
Device: TMS fMRI — compare measurements to established functional connectivity measures; e.g., EEG coherence and fMRI

SUMMARY:
Background:

People tend to pay more attention to one side of space than the other and this may be due to differences in the structure and function of the two sides of the brain. We are interested in whether we can detect those difference with magnetic resonance imaging (MRI), transcranial magnetic stimulation (TMS), and electroencephalography (EEG).

Objective:

The purpose of the study is to understand how differences in brain structure may cause people to pay more attention to one side than the other.

Eligibility:

Healthy adults ages 18-35

Design:

Participants will be screened with a neurological exam.

Participants will have 2-3 visits for a total duration of about 7/8 hours.

Women of childbearing age must have a negative pregnancy test before each MRI scan.

Visits may include:

Physical exam

Tests of attention, and thinking

TMS. A brief electrical current will pass through a wire coil on the scalp. Participants will hear a click and may feel a pull. They may be asked to tense muscles or do tasks.

Magnetic resonance imaging (MRI) scan for a maximum of 1 hour. Participants will lie on a table that slides into a cylinder in a strong magnetic field. They will do tasks on a computer screen or lie still. They will get earplugs for loud noise.

EEG for no longer than 5 hours, with most lasting 3 hours. Gel and a cap with electrodes will be placed on the scalp. They will record brain waves while the participant gets TMS or does nothing.

Questions about participants dominant hand and about the MRI.

DETAILED DESCRIPTION:
Objective

The goal of this protocol to explore correlations between lateralized individual differences in visual attentional preference and hemispheric asymmetries in functional connectivity between the frontal and parietal visual attention areas. To measure functional connectivity, resting state functional MRI and electroencephalographic (EEG) potentials evoked with transcranial magnetic stimulation (TMS) will be used. Protocol research will also attempt to validate the TMS-evoked EEG potentials against fMRI resting state functional connectivity.

Study Population

Up to 80 right-handed and right-eyed healthy volunteers, aged 18-35

Design

TMS evoked EEG potentials (TEPs) and fMRI will be used to measure functional connectivity between the posterior parietal cortex and the frontal visual attention area. Various tasks will be used to quantify attention and explore their relationship with asymmetries in functional connectivity. A qualitative comparison between the value of fMRI and TEPs for predicting attentional bias will be made.

Outcome Measures

* Behavioral measures of attention
* TEP measures of functional connectivity
* fMRI measures of functional connectivity

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age 18 and older
* Able to provide consent

For some sub-studies, we may limit participation by handedness or eye dominance.

EXCLUSION CRITERIA:

* Any current major neurological or psychiatric disorder, such as, (but not limited to) stroke, Parkinson disease, Alzheimer disease, schizophrenia or major depression
* Findings on neurological examination indicative of significant brain disease
* Individuals with significant health problems, such as cardiovascular disease, malignancy, or connective tissue disorder
* History of seizure, defined as a diagnosis by a health care provider of one or more epileptic seizures or an anecdotal history which, in the opinion of the PI, is suggestive of epileptic seizure. Any individual who answers other than negatively to the question, Have you ever had an epileptic seizure on screening will be questioned directly by the PI
* Current oral use of a medication that lowers the seizure threshold such as neuroleptics, beta lactams, isoniazid, metronidazole, tricyclic or other antidepressants, or prescription stimulants
* Individuals regularly taking medications that cause significant psychomotor activation or depression, e.g., stimulants and CNS depressant drugs such as benzodiazepines, will be excluded.
* For MRI studies: Any metal in the body which would make having an MRI scan unsafe, such as pacemakers, stimulators, pumps, aneurysm clips, metallic prostheses, artificial heart valves, cochlear implants or shrapnel fragments, any individual who was a welder or metal worker. Participants will also be excluded if they are uncomfortable in small closed spaces (i.e. claustrophobia) or are not able to lie comfortably on their back for up to two hours
* Pregnancy or plans to become pregnant in the next two months
* Members of the Behavioral Neurology Unit, NINDS
* Use of illegal drugs in the past year
* Consumption of more than 7 alcoholic drinks a week for females or 14 alcoholic drinks a week for males.

There is no general exclusion for NIH employees. Inclusion/exclusion criteria will be checked before enrollment in each sub-study to ensure that participants remain eligible.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2022-10-24 (Actual)

PRIMARY OUTCOMES:
Exploratory sub-studies under this protocol will answer questions about how to optimize EEG recordings of the cortical response to TMS. | 20 visits
  Response to TMS

CONTACTS AND LOCATIONS:
Overall Officials: Eric M Wassermann, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
.Data sharing at an independent subject level may not be feasible.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2019-N-0036.html